CLINICAL TRIAL: NCT04026750
Title: A Randomized, Double-Blind, Placebo-Controlled Insulin Tolerance Test Study to Assess the Safety, Tolerability, and Pharmacodynamics OF Pitolisant in Patients With Type 1 Diabetes
Brief Title: Insulin Tolerance Test Study in Patients With Type 1 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on scientific data collected during the trial and high screen fail rate.
Sponsor: High Point Clinical Trials Center (Industry)
Collaborators: Ferox Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FPITO-T1D-01.01
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pitolisant (Experimental)
  Interventions: Drug: Pitolisant
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Pitolisant

INTERVENTIONS:
Drug: Pitolisant — Pitolisant will be administered orally for 7 days. Patients may have their study drug dose adjusted downward if the starting dose is not tolerated.

SUMMARY:
The primary objective of this study is to determine the safety, tolerability and pharmacodynamics of pitolisant in patients with Type 1 Diabetes

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Diagnosis of diabetes => 4yrs, On Insulin => 4yrs, HbA1c<= 10%, At least one episode of severe hypoglycemia in past 12 months, fasting c-peptide <0.7 ng/ml

Exclusion Criteria:

* Hypoglycemia unawareness, DKA within 3 months prior to randomization, Reduced renal function, Anxiety and depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Fein, MD, Principal Investigator — PI
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pitolisant 36mg: 2-18mg tablets once daily for 7 days
- Placebo: 2- Placebo tablets to match pitolisant 18mg once daily for 7 days
Period: Overall Study
Arm/Group | Pitolisant 36mg | Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pitolisant 36mg: 2-18 mg tablets per day for 7 days
- Placebo: 2-Placebo to match 18mg of pitolisant
- Total: Total of all reporting groups
Arm/Group | Pitolisant 36mg | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (5.57) | 43.5 (12.02) | 36.6 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Glucagon Response to Hypoglycemia
Description: Change in peak glucagon concentration from day 1 ITT (baseline) to day 7 ITT (on treatment). Serial glucagon collected during ITT's, occurred at -10, 0, 15, 30, 45, 60, 90, 120 and 180 minutes just prior to and during the ITT.
Time Frame: Change in peak glucagon during ITT Day 1 vs. Day 7
Measure: Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Placebo: 2- Placebo to match pitolisant 18mg once daily for 7 days
Arm/Group | Pitolisant 36mg | Placebo
Number analyzed (Participants) | 3 | 2
pg/mL | 7.5 [-2.07 to 17.02] | 13.1 [2.08 to 24.07]

2. Secondary Outcome: Number of Patients Returning to Blood Glucose =>70 mg/dL
Description: Number of patients that returned to blood glucose =>70 mg/dL during ITT
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 2- Placebo to match pitolisant once daily for 7 days
Arm/Group | Pitolisant 36mg | Placebo
Number analyzed (Participants) | 3 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to day 16
Arm/Group | Pitolisant 36mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pitolisant 36mg (N=3) | Placebo (N=2)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (55) | 2 (86) — Blood Glucose < 70 mg/dL
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04026750/Prot_SAP_000.pdf